CLINICAL TRIAL: NCT06526793
Title: A Modular Phase 2, Single-arm, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Surovatamig (AZD0486) in Participants With Relapsed or Refractory (R/R) B-cell Non-Hodgkin Lymphoma (SOUNDTRACK-B)
Brief Title: Surovatamig (AZD0486) as Monotherapy in Participants With Relapsed/Refractory (R/R) B-cell NHL
Acronym: SOUNDTRACK-B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7404C00001; 2023-505789-27-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-07-03; First posted 2024-07-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: B-cell Non-Hodgkin Lymphoma; Follicular Lymphoma (FL); Large B-Cell Lymphoma (LBCL)
Keywords: AZD0486; Surovatamig; Follicular Lymphoma (FL); Large B-Cell Lymphoma (LBCL); Non-Hodgkin lymphoma (NHL); Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Recurrence

STUDY DESIGN:
Intervention Model Description: The trial will assess surovatamig (AZD0486) monotherapy given by IV infusion. Module 1 will evaluate the efficacy and safety of surovatamig monotherapy at the recommended Phase 2 dose (RP2D), in participants 18 years of age or older , with relapsed or refractory (R/R) follicular lymphoma (FL) who have received ≥ 2 prior therapies. Module 2 will evaluate the efficacy and safety of surovatamig monotherapy at the RP2D for participants 18 years of age or older with (R/R) large B-cell lymphoma (LBCL) who have received ≥ 2 prior therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1: Surovatamig Monotherapy in Participants with Relapsed or Refractory Follicular Lymphoma (Experimental): In Module 1, the efficacy and safety of surovatamig at the RP2D will be evaluated in R/R FL. Surovatamig will be administered as intravenous infusion.
  Interventions: Drug: Surovatamig
- Module 2: Surovatamig Monotherapy in Participants with Relapsed or Refractory LBCL (Experimental): In Module 2, the efficacy and safety of surovatamig at the RP2D will be evaluated in R/R LBCL. Surovatamig will be administered as intravenous infusion.
  Interventions: Drug: Surovatamig

INTERVENTIONS:
Drug: Surovatamig — Investigational Product administered via intravenous infusion.
  Other Names: AZD0486

SUMMARY:
This is a Phase 2 global, multi-center, open-label study to assess the efficacy, safety and tolerability of Surovatamig (AZD0486) monotherapy in adult participants with relapsed/refractory B-cell non-Hodgkin lymphoma (NHL) who have received at least two prior lines of therapies. The study has 2 Modules: Module 1 for FL and Module 2 for LBCL.

DETAILED DESCRIPTION:
This is a modular, Phase II, multicenter, single-arm, open-label study to evaluate the efficacy and safety of Surovatamig (AZD0486) monotherapy administered as an intravenous (IV) infusion in participants with relapsed or refractory B-NHL. The purpose of this study is to determine the efficacy and safety of AZD0486 administered at the RP2D in adults 18 years of age or older with relapsed or refractory B-NHL.

ELIGIBILITY:
1. Key Inclusion Criteria:

   * Aged 18 years old and above
   * Histologically confirmed relapsed refractory FL (Module 1) and LBCL (Module 2) after at least 2 prior lines of therapy
   * ECOG performance status 0 to 2
   * Locally confirmed CD-19 expression in lymphoma cells after progression from last CD 19 directed therapy
   * FDG-avid disease with at least one bi-dimensionally measurable nodal lesion (defined as > 1.5 cm in its longest dimension), or extranodal lesion (defined as > 1.0 cm in its longest dimension)
   * Adequate hematological function: ANC ≥ 1000/mm3, platelets

     * 75,000/mm3, hemoglobin ≥ 9 g/dL. Transfusion and/or growth factor are allowed but counts must be stable for at least 72 hours afterwards prior to screening
   * Adequate liver function: total bilirubin <1.5x ULN, AST/ALT ≤ 3xULN or < 5 × ULN in the presence of lymphoma involvement of the liver
   * Adequate renal function: creatinine clearance (CrCl) of ≥ 45 mL/min
   * Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) ≥ 45% by echocardiogram or MUGA

   The above is a summary, other inclusion criteria details may apply.
2. Key Exclusion Criteria:

   * Diagnosis of CLL, Burkitt lymphoma, or Richter's transformation
   * Active CNS involvement by B-NHL
   * Leukemic presentation of B-NHL
   * History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, neurodegenerative disorder including Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis or other severe mental illness
   * Prior therapy with T-cell engager (TCE) within 8 weeks, autologous Hematopoietic Stem Cell Transplantation (HSCT) within 12 weeks, CAR T- cell therapy within 6 months, or prior allogeneic HSCT within 24 weeks of first dose of surovatamig
   * Requires chronic immunosuppressive therapy
   * Unresolved non hematological AEs ≥ Grade 2 from prior therapies; history of ≥ Grade 3 CRS or neurotoxicity from prior CAR-T or TCE therapy
   * History of major cardiac abnormalities.
   * If female, participant must not be pregnant or breastfeeding.

The above is a summary, other exclusion criteria details may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2029-06-14 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (central review) | Module 1: from first dose to end of treatment or data cutoff, whichever comes first, assessed up to approximately 24 months. Module 2: from first dose to end of treatment or data cutoff, whichever comes first, assessed up to approximately 12 months.
  Overall response rate (ORR), defined as the proportion of participants achieving either a Partial Response (PR) or Complete Response (CR) based on Lugano 2014 response criteria for non-Hodgkin Lymphoma, as determined by central review

SECONDARY OUTCOMES:
Incidence, nature and severity of Adverse Events (AEs), Serious AEs and AEs of Special Interest (AESI) | From time of Informed Consent to 90-day safety follow-up visit
  Incidence, nature, and severity of AEs/SAEs (based on NCI CTCAE v5.0/ASTCT criteria/Cairo-Bishop criteria with Howard modification) and changes in laboratory data, vital signs, and electrocardiograms (ECGs) compared with baseline.
  Incidence and severity of AESIs.
Incidence and nature of study drug discontinuation, dose reduction, and dose delay due to Adverse Events (AEs) | From the start of treatment up to 2 years in Module 1 and up to 1 year for Module 2
  Incidence and nature of study drug discontinuation, dose reduction, and dose delay due to AEs
Duration of response (DoR) | To be assessed up to approximately 5 years.
  Defined as the time from the date of first documented response until date of documented progression by Lugano 2014 response criteria as determined by central review or death due to any cause.
Complete response (CR) rate (central review) | To be assessed up through study completion, up to approximately 5 years
  Complete response (CR) based on Lugano 2014 Response criteria for non-Hodgkin lymphoma, as determined by central review.
Complete response (CR) rate (investigator assessment) | To be assessed up through study completion, up to approximately 5 years
  Complete response (CR) based on Lugano 2014 Response criteria of non-Hodgkin lymphoma, as determined by investigator assessment.
Overall response rate (ORR) (investigator assessment) | Module 1: from first dose to end of treatment or data cutoff, whichever comes first, assessed up to about 24 months. Module 2: from first dose to end of treatment or data cutoff, whichever comes first, assessed up to about 12 months.
  Overall response rate (ORR), defined as the proportion of participants achieving either a partial response (PR) or complete response (CR) based on Lugano 2014 Response criteria of non-Hodgkin lymphoma, as determined by investigator assessment.
Duration of complete response (DoCR) | To be assessed up to approximately 5 years.
  Defined as the time from achievement of complete response (CR) to relapse or death due any cause, as assessed by central review
Time to response (TTR) | From the first dose until the first objective response, up to approximately 5 years.
  Defined as the time from first dose until first documented objective response, as assessed by central review.
Event-free survival (EFS) | To be assessed up to approximately 5 years
  Defined as the time from first dose until disease progression, relapse, or initiation of subsequent systemic anti-lymphoma treatment, or death due to any cause, as assessed by central review.
Progression-free survival (PFS) | To be assessed up to approximately 5 years.
  Defined as the time from the date of first dose until documented disease progression based on Lugano 2014 Response Criteria, or death due to any cause.
Time to next anti-lymphoma (TTNT) | To be assessed up to approximately 5 years.
  Defined as time from first dose until the start of subsequent anti-lymphoma therapy.
Overall survival (OS) | To be assessed up to approximately 5 years.
  Defined as the time from first dose until the date of death due to any cause.
Plasma concentrations of surovatamig | From Cycle 1 Day 1 (pre-dose) (each cycle is 28 days) up to 90 days after end of treatment
  To characterize the plasma concentration of surovatamig as monotherapy
Area under the concentration time curve (AUC) | From Cycle 1 Day 1 (pre-dose) (each cycle is 28 days) up to 90 days after end of treatment
  To characterize the pharmacokinetics (PK) AUC of surovatamig as monotherapy
Maximum plasma concentration (Cmax) | From Cycle 1 Day 1 (pre-dose) (each cycle is 28 days) up to 90 days after end of treatment
  To characterize the pharmacokinetics (PK) (Cmax) of surovatamig as monotherapy
Time to maximum plasma concentration (Tmax) | From Cycle 1 Day 1 (pre-dose) (each cycle is 28 days) up to 90 days after end of treatment
  To characterize the pharmacokinetics (PK) (Tmax) of surovatamig as monotherapy
A trough concentration (Cthrough) | From Cycle 1 Day 1 (pre-dose) (each cycle is 28 days) up to 90 days after end of treatment
  To characterize the pharmacokinetics (PK) (C through) of surovatamig as monotherapy
Immunogenecity of surovatamig | From the first dose of study intervention, at predefined intervals throughout the administration of surovatamig (2 years in Module 1 and 1 year in Module 2)
  The number and percentage of participants who develop Anti-Drug Antibodies (ADAs)
Change from baseline in EORTC IL233 scales | To be assessed up through study completion, up to approximately 5 years
  To evaluate patient-reported tolerability of surovatamig, including severity of key treatment-related symptoms and overall side-effect burden
  EORCT IL233 scales - European Organisation for Research and Treatment of Cancer Il233 scales- this questionnaire is assessing Patient-reported Severity of Treatment-and Disease-related Symptoms, it is a 15-item questionnaire, and each item is rated on a 4-point scale ranging from 1 (not at all) to 4 (very much).
Change from baseline in PGI-T scale | To be assessed up through study completion, up to approximately 5 years
  To evaluate patient-reported tolerability of surovatamig, overall side-effect burden.
  PGI-T scale - Patient Global Impression of Treatment Tolerability is a 1 item questionnaire rated on a 7-point scale ranging from "not at all" to "very much"
Change from baseline in EORTC IL 232 QL2 scores | To be assessed up through study completion, up to approximately 5 years
  To evaluate patient-reported severity of key disease-related symptoms, as well as the impact of disease on lymphoma-specific concerns, while on surovatamig.
  European Organization for Research and Treatment of Cancer (EORTC) IL 232 will be used to evaluate impacts on function and HRQoL due to treatment and disease, which includes 13 EORTC QLQ-C30 function items assessing physical, social, role, and emotional function, as well as the EORTC QLQ-C30's 2 global health/HRQoL items.
Change from baseline in FACT-LymS scales | To be assessed up through study completion, up to approximately 5 years
  To evaluate patient-reported severity of key disease-related symptoms, as well as the impact of disease on lymphoma-specific concerns, while on surovatamig
  Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) FACT-LymS - Lymphoma-specific Subscale from the FACT-Lym Questionnaire is a 15-item questionnaire, and each item is rated on a 5-point scale ranging from 0 (not at all) to 4 (very much).
Minimal residual disease (MRD) | To be assessed up through study completion, up to approximately 5 years
  MRD-negative complete response (CR) rate, defined as the proportion of participants who achieved MRD-negativity in plasma by next generation sequencing (NGS) while in complete response (CR) per the Lugano Response criteria for non-Hodgkin lymphoma as determined by central review.

CONTACTS AND LOCATIONS:
Locations (83):
- United States (22):
  - Research Site, Phoenix, Arizona
  - Research Site, Duarte, California
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Waukee, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (4):
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Macquarie University
  - Research Site, Nedlands
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (4):
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- China (9):
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Zhengzhou
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Vejle
- France (4):
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Rouen
- Germany (5):
  - Research Site, Berlin
  - Research Site, Chemnitz
  - Research Site, Essen
  - Research Site, Jena
  - Research Site, Würzburg
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Italy (5):
  - Research Site, Alessandria
  - Research Site, Bologna
  - Research Site, Busto Arsizio
  - Research Site, Milan
  - Research Site, Roma
- Japan (8):
  - Research Site, Chiba
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Yokohama
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pozuelo de Alarcón
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (5):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements: thttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://vivli.org/